CLINICAL TRIAL: NCT07268872
Title: Dynamic Effects of Different Anesthetic Agents on the Immune Function of Healthy Volunteers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HenanPPH-LFF
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Immune System
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propofol group (Active Comparator): Anesthesia induction: 1.5-2.5 mg/kg IV bolus; Anesthesia maintenance: 4-12 mg/kg/h infusion
  Interventions: Drug: Propofol group
- Sevoflurane group (Active Comparator): Anesthesia induction: 6% concentration inhaled for 2 minutes; Anesthesia maintenance: 0.5-3% concentration
  Interventions: Drug: Sevoflurane group
- Ciprofol group (Active Comparator): Anesthesia induction: 0.4 mg/kg IV injection over 10-30s; if anesthesia depth is insufficient, additional doses not exceeding 0.2 mg/kg may be given; Anesthesia maintenance: 0.4-2.4 mg/kg/h infusion
  Interventions: Drug: Ciprofol group
- Control group (Placebo Comparator): subjects will not undergo anesthesia but will remain in a supine position on a hospital trolley for 3 hours.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Propofol group — Induction with 1.5-2.5 mg/kg IV bolus until loss of consciousness (loss of eyelash reflex), maintenance with 4-12 mg/kg/h target-controlled infusion.
  Arms: Propofol group
Drug: Sevoflurane group — Induction with 8% concentration inhaled for approximately 2 minutes, maintenance concentration 0.5-3%.
  Arms: Sevoflurane group
Drug: Ciprofol group — Induction with 0.4 mg/kg IV bolus over 10-30s; if anesthesia depth is insufficient, additional doses not exceeding 0.2 mg/kg may be given; maintenance with 0.4-2.4 mg/kg/h target-controlled infusion.
  Arms: Ciprofol group
Other: Control group — subjects will not receive anesthesia but will remain in a supine position on a hospital trolley for 3 hours, after which they will be sent to the Post-Anesthesia Care Unit (PACU).
  Arms: Control group

SUMMARY:
This study recruits healthy volunteers and randomly assigns them in a 1:1:1:1 ratio to the following groups: Propofol group, Sevoflurane group, Ciprofol group, and Control group. Subjects in the different groups will undergo anesthesia with the corresponding general anesthetic drug, while subjects in the Control group will receive no anesthesia. Peripheral blood samples will be collected at specified time points: before anesthesia induction, upon emergence from anesthesia, 24 hours after anesthesia, and 48 hours after anesthesia. Single-cell multi-omics analysis will be performed on these samples using single-cell sequencing technology. The aim is to investigate the independent effects of different general anesthetic drugs on human immune function in the absence of surgical trauma, and to further explore the potential immunomodulatory effects of commonly used clinical anesthetics.

ELIGIBILITY:
Inclusion Criteria:

Volunteers undergo routine blood tests, liver function, kidney function, coagulation function, and routine 12-lead electrocardiogram examination before the trial. Any item showing no significant abnormalities; Age 20-30 years; ASA physical status I; BMI (Body Mass Index) 18-28 kg/m².

Exclusion Criteria:

History of neurological/psychiatric diseases, immune system diseases, or any type of chronic disease; History of surgical anesthesia; History of bad habits such as drug abuse, smoking or excessive drinking; Women during menstruation, pregnancy, or lactation; Recent use of immunosuppressants, hormones, non-steroidal anti-inflammatory drugs; Intake of antibiotics, probiotics, prebiotics, or other supplements within three months prior to stool sample collection; Recent history of diarrhea, inflammatory bowel disease, or other diseases severely affecting gut microbiota structure.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Single-cell multi-omics data obtained from peripheral blood mononuclear cells; metabolome, lipidome, and proteome data obtained from plasma through detection; whole genome sequencing data. | Peripheral blood samples will be collected at specified time points: before anesthesia induction, upon emergence from anesthesia, 24 hours after anesthesia, and 48 hours after anesthesia. Single-cell multi-omics analysis will be performed on these sample

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial People's Hospital, Henan, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No